CLINICAL TRIAL: NCT01691534
Title: A Phase 2 Trial to Evaluate the Early Bactericidal Activity, Safety and Tolerability of the Following: TMC207 Plus PA-824 Plus Pyrazinamide Plus Clofazimine, TMC207 Plus PA-824 Plus Pyrazinamide, TMC207 Plus PA-824 Plus Clofazimine Alone, TMC207 Plus Pyrazinamide Plus Clofazimine, Pyrazinamide Alone, and Clofazimine Alone; in Adult Patients With Newly Diagnosed, Smear-Positive Pulmonary Tuberculosis.
Brief Title: Evaluation of Early Bactericidal Activity in Pulmonary Tuberculosis With Clofazimine (C)-TMC207 (J)-PA-824 (Pa)-Pyrazinamide (Z)
Acronym: NC-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NC-003-(C-J-Pa-Z)
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; EBA; PA824; pretomanid; TMC207
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — bedaquiline; pretomanid; Pyrazinamide; Clofazimine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- TMC207, PA-824, pyrazinamide and clofazimine (J-PA-Z-C) (Experimental): TMC207 400 mg Day 1; 300mg Day 2; 200mg Days 3-14 plus PA-824 200mg Days 1-14 plus pyrazinamide 1500mg Days 1-14 plus clofazimine 300mg Days 1-3 and Clofazamine 100mg Days 4-14
  Interventions: Drug: TMC207 (J); Drug: PA-824 (PA); Drug: pyrazinamide (Z); Drug: clofazimine (C)
- TMC207, PA-824 and pyrazinamide (J-PA-Z) (Experimental): TMC207 400 mg Day 1; 300mg Day 2; 200mg Days 3-14 plus PA-824 200mg Days 1-14 plus pyrazinamide 1500mg Days 1-14
  Interventions: Drug: TMC207 (J); Drug: PA-824 (PA); Drug: pyrazinamide (Z)
- TMC207, PA-824 and clofazimine (J-PA-C) (Experimental): TMC207 400 mg Day 1; 300mg Day 2; 200mg Days 3-14 plus PA-824 200mg Days 1-14 plus clofazimine 300mg Days 1-3 and clofazimine 100mg Days 4-14
  Interventions: Drug: TMC207 (J); Drug: PA-824 (PA); Drug: clofazimine (C)
- TMC207, pyrazinamide and clofazimine (J-Z-C) (Experimental): TMC207 400 mg Day 1; 300mg Day 2; 200mg Days 3-14 plus pyrazinamide 1500mg Days 1-14 plus clofazimine 300mg Days 1-3 and Clofazimine 100mg Days 4-14
  Interventions: Drug: TMC207 (J); Drug: pyrazinamide (Z); Drug: clofazimine (C)
- pyrazinamide (Z) (Experimental): pyrazinamide 1500mg Days 1-14
  Interventions: Drug: pyrazinamide (Z)
- clofazimine (C) (Experimental): Clofazimine 300mg Days 1-3 and Clofazimine 100mg Days 4-14
  Interventions: Drug: clofazimine (C)
- Rifafour (Active Comparator): Rifafour e-275 mg dosed by weight
  Interventions: Drug: Rifafour

INTERVENTIONS:
Drug: TMC207 (J) — TMC207 400 mg Day 1; 300mg Day 2; 200mg Days 3-14
  Arms: TMC207, PA-824 and clofazimine (J-PA-C); TMC207, PA-824 and pyrazinamide (J-PA-Z); TMC207, PA-824, pyrazinamide and clofazimine (J-PA-Z-C); TMC207, pyrazinamide and clofazimine (J-Z-C)
Drug: PA-824 (PA) — PA-824 200mg Days 1-14
  Arms: TMC207, PA-824 and clofazimine (J-PA-C); TMC207, PA-824 and pyrazinamide (J-PA-Z); TMC207, PA-824, pyrazinamide and clofazimine (J-PA-Z-C)
Drug: pyrazinamide (Z) — 1500mg Days 1-14 Dosed by Weight
  Arms: TMC207, PA-824 and pyrazinamide (J-PA-Z); TMC207, PA-824, pyrazinamide and clofazimine (J-PA-Z-C); TMC207, pyrazinamide and clofazimine (J-Z-C); pyrazinamide (Z)
Drug: clofazimine (C) — clofazimine 300mg Days 1-3 and clofazimine 100mg Days 4-14
  Arms: TMC207, PA-824 and clofazimine (J-PA-C); TMC207, PA-824, pyrazinamide and clofazimine (J-PA-Z-C); TMC207, pyrazinamide and clofazimine (J-Z-C); clofazimine (C)
Drug: Rifafour — Rifafour e-275 mg dosed by weight
  Arms: Rifafour

SUMMARY:
The trial will evaluate the extended bactericidal activity of 14 consecutive days of oral administration of TMC207 plus PA-824 plus Pyrazinamide plus Clofazimine, TMC207 plus PA-824 plus Pyrazinamide, TMC207 plus PA-824 plus Clofazimine alone, TMC207 plus Pyrazinamide plus Clofazimine, Pyrazinamide alone, Clofazimine alone, and standard first line TB treatment as per South African TB Guidelines (Rifafour e-275) as determined by the rate of change of log CFU per ml sputum over the time period Day 0-14 in participants with smear positive pulmonary tuberculosis (TB). A control group will receive standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provide written, informed consent prior to all trial-related procedures including HIV testing.

  2. Male or female, aged between 18 and 65 years inclusive.

  3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.

  4. Newly diagnosed, previously untreated, sputum smear-positive pulmonary TB.

  5. A chest X-ray picture which in the opinion of the Investigator is compatible with TB.

  6. Sputum positive GeneXpert or TB Smear from TB clinic or site initial diagnosis

  7. Sputum positive on direct microscopy for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale).

  8. Ability to produce an adequate volume of sputum as estimated from a spot assessment (estimated 10 ml or more overnight production).

  9. Be of non-childbearing potential or using an effective method of birth control as defined as:

Non-childbearing potential:

1. Subject - Not heterosexually active or practice sexual abstinence or
2. Female subject/sexual bilateral oophorectomy, bilateral tubal ligation, and/or hysterectomy or has been postmenopausal with a history of no menses for at least 12 consecutive months) or
3. Male subject/sexual partner - vasectomised or has had a bilateral orchidectomy minimally three month prior to screening

Effective birth control methods:

1. Double barrier method which can include a male condom, diaphragms, cervical cap, or female condom or
2. Barrier method combined with hormone based contraceptives or an intra-uterine device for the female partner and are willing to continue practicing birth control methods throughout treatment and for 12 weeks (male participants) or 6 months (female participants) after the last dose of study medication or discontinuation from study medication in case of premature discontinuation

(Note: Hormone-based contraception alone may not be reliable when taking IMP; therefore, hormone-based contraceptives alone cannot be used by female participants to prevent pregnancy).

Exclusion Criteria:

1. Evidence of clinically significant (as judged by the investigator), metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied) including malaria.
2. Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
3. A history of previous TB.
4. Clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
5. History of allergy to the IMP or related substances.
6. Isoniazid-resistant and/or Rifampicin-resistant bacteria detected with a sputum specimen collected within the pre-treatment period and tested at the study laboratory.
7. Known or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the participant.
8. HIV infected participants:

   1. having a CD4+ count <200 cells/µL;
   2. or having received antiretroviral therapy medication within the last 90 days;
   3. or having received oral or intravenous antifungal medication within the last 90 days;
   4. or with an AIDS-defining opportunistic infection or malignancies (except pulmonary TB).
9. Having participated in other clinical studies with investigational agents within 8 weeks prior to trial start.
10. Significant cardiac arrhythmia requiring medication.
11. Participants with the following at screening. For ECGs, central cardiology overread and the mean of triplicate reading must be used:

    1. Marked prolongation of QT/QTc interval, e.g., confirmed demonstration of QTcF (Fridericia correction) or QTcB (Bazett correction) interval >450 ms at screening;
    2. History of additional risk factors for Torsade de Pointes, e.g., heart failure, hypokalemia, family history of Long QT Syndrome;
    3. Use of concomitant medications that prolong the QT/QTc interval (see exclusion criterion 19 and disallowed medications;
    4. Pathological Q waves (defined as >40ms or depth >0.4-0.5mV);
    5. ECG evidence of ventricular pre-excitation;
    6. ECG evidence of complete or incomplete left bundle branch block or right bundle branch block;
    7. ECG evidence of second or third degree heart block;
    8. Intraventricular conduction delay with QRS duration >120ms;
    9. Bradycardia as defined by sinus rate <50bpm.
12. Females who are pregnant, breast-feeding, or planning to conceive a child within 6 months of cessation of treatment. Males planning to conceive a child within twelve weeks of cessation of treatment.
13. Diabetes Mellitus requiring insulin.
14. History of lens opacity.
15. For males, any history of a clinically significant abnormality in the reproductive system.

    Specific Treatments
16. Previously received treatment with Clofazimine, TMC207 or PA-824.
17. Treatment received with any drug active against MTB within the 3 months prior to Visit 1 (e.g. isoniazid, ethambutol, amikacin, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides, metronidazole).
18. Any diseases or conditions in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to allergy to any TB drug, their component or to the IMP.
19. Concomitant use of any drug known to prolong QTc interval (including amiodarone, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, cyclobenzaprine, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, thioridazine).
20. Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes (such as quinidine, tyramine, ketoconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan). Exceptions may be made for participants that have received 3 days or less of one of these drugs or substances, if there has been a wash-out period before administration of IMP equivalent to at least 5 half-lives of that drug or substance.
21. Use of any therapeutic agents known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine) within 30 days prior to dosing. Exceptions for opiate and pain killer use for cough or underlying disease may be made at investigator discretion.

    Based on Laboratory Abnormalities
22. Participants with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (November 2007):

    1. creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]);
    2. lipase grade 3 or greater (>2.0 x ULN);
    3. hemoglobin grade 4 (<6.5 g/dL);
    4. platelets grade 2 or greater (under 50x109 cells/L);
    5. serum potassium grade 2 or greater (<3.5 mEq/L);
    6. aspartate aminotransferase (AST) grade 3 (≥3.0 x ULN) to be excluded;
    7. alanine aminotransferase (ALT) grade 3 (≥3.0 x ULN) to be excluded;
    8. alkaline phosphatase (ALP) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 x ULN) must be discussed with the sponsor Medical Monitor;
    9. total bilirubin grade 3 or greater (>2.0 x ULN, or >1.50 x ULN when accompanied by any increase in other liver function test) to be excluded, grade 2 (>1.50 x ULN, or >1.25 x ULN when accompanied by any increase in other liver function test) must be discussed with the sponsor Medical Monitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Diacon, MD, Principal Investigator — Karl Bremer Hospital, Cape Town South Africa
Locations (2):
- South Africa (2):
  - Centre for Tuberculosis Research Innovation, UCT Lung Institute, Cape Town
  - Task Applied Science, Karl Bremer Hospita, Cape Town

REFERENCES:
- [Derived] Diacon AH, Dawson R, von Groote-Bidlingmaier F, Symons G, Venter A, Donald PR, van Niekerk C, Everitt D, Hutchings J, Burger DA, Schall R, Mendel CM. Bactericidal activity of pyrazinamide and clofazimine alone and in combinations with pretomanid and bedaquiline. Am J Respir Crit Care Med. 2015 Apr 15;191(8):943-53. doi: 10.1164/rccm.201410-1801OC. PMID 25622149

RESULTS

PARTICIPANT FLOW:
Groups:
- TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C): TMC207 (J): 400 mg on Day 1; 300 mg on Day 2; and 200 mg on Days 3 to 14
  PA-824 (PA): 200 mg on Days 1 to 14
  pyrazinamide (Z): 1500 mg on Days 1 to 14
  clofazimine (C): 300 mg on Days 1 to 3 and 100 mg on Days 4-14
- TMC207, PA-824 and Pyrazinamide (J-PA-Z): TMC207 (J): 400 mg on Day 1; 300 mg on Day 2; and 200 mg on Days 3 to 14
  PA-824 (PA): 200 mg on Days 1 to 14
  pyrazinamide (Z): 1500 mg on Days 1 to 14
- TMC207, PA-824 and Clofazimine (J-PA-C): TMC207 (J): 400 mg on Day 1; 300 mg on Day 2; and 200 mg on Days 3 to 14
  PA-824 (PA): 200 mg on Days 1 to 14
  clofazimine (C): 300 mg on Days 1 to 3 and 100 mg on Days 4-14
- TMC207, Pyrazinamide and Clofazimine (J-Z-C): TMC207 (J): 400 mg on Day 1; 300 mg on Day 2; and 200 mg on Days 3 to 14
  pyrazinamide (Z): 1500 mg on Days 1 to 14
  clofazimine (C): 300 mg on Days 1 to 3 and 100 mg on Days 4-14
- Pyrazinamide (Z): pyrazinamide (Z): 1500 mg on Days 1 to 14
- Clofazimine (C): clofazimine (C): 300 mg on Days 1 to 3 and 100 mg on Days 4-14
- Rifafour: Rifafour on Days 1 to 14, dosed by weight
Period: Overall Study
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Started | 15 | 15 | 15 | 15 | 15 | 15 | 15
Completed | 15 | 14 | 14 | 14 | 15 | 14 | 14
Not Completed | 0 | 1 | 1 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.74) | 33.4 (14.22) | 33.3 (11.15) | 30.9 (13.12) | 32.4 (11.44) | 28.4 (8.77) | 34.3 (10.25) | 32.6 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 8 | 6 | 6 | 6 | 8 | 40
  Male | 12 | 12 | 7 | 9 | 9 | 9 | 7 | 65
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 9 | 5 | 6 | 8 | 8 | 6 | 9 | 51
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Mixed Ethnic | 6 | 9 | 9 | 7 | 6 | 9 | 6 | 52
Height [Mean (Standard Deviation); unit: centimeters] | 168.6 (7.98) | 165.3 (8.64) | 166.8 (11.37) | 166.6 (11.86) | 165.1 (7.58) | 167.8 (9.05) | 164.3 (8.74) | 166.3 (9.28)
Weight [Mean (Standard Deviation); unit: kilograms] | 56.4 (9.49) | 50.2 (7.36) | 57.4 (10.58) | 58.7 (9.21) | 52.4 (7.21) | 53.3 (9.41) | 56.1 (10.80) | 55.0 (9.43)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 19.9 (3.66) | 18.4 (1.98) | 21.0 (4.64) | 21.3 (3.34) | 19.2 (1.86) | 18.8 (2.15) | 20.8 (3.29) | 19.9 (3.23)
HIV Status [Number; unit: participants]
  Negative | 14 | 14 | 12 | 15 | 13 | 14 | 11 | 93
  Doubtful | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Positive | 1 | 1 | 3 | 0 | 2 | 1 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Early Bactericidal Activity (EBA) Measured as the Daily Rate of Change in log10 CFUs (Colony Forming Units) of M. Tuberculosis in Sputum on Solid Media (Days 0-14).
Time Frame: 14 consecutive days of treatment
Population: Efficacy population: all patients included in the safety population for whom corresponding efficacy data were available and had no major protocol violations/deviations defined as protocol violations/deviations affecting the integrity of the efficacy data
Measure: Mean (95% Confidence Interval); unit: log10CFU/ml/day
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Number analyzed (Participants) | 13 | 12 | 15 | 13 | 15 | 14 | 15
log10CFU/ml/day | 0.115 [0.039 to 0.189] | 0.167 [0.075 to 0.257] | 0.076 [0.005 to 0.145] | 0.124 [0.035 to 0.214] | 0.036 [-0.026 to 0.099] | -0.017 [-0.085 to 0.053] | 0.151 [0.071 to 0.232]

2. Secondary Outcome: EBA Measured as the Daily Rate of Change in log10 CFUs of M. Tuberculosis in Sputum on Solid Media (Days 0-2)
Time Frame: Days 0-2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: log10CFU/ml/day
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Number analyzed (Participants) | 13 | 12 | 15 | 13 | 15 | 14 | 15
log10CFU/ml/day | 0.161 [0.042 to 0.279] | 0.196 [0.061 to 0.330] | 0.062 [-0.045 to 0.161] | 0.132 [0.008 to 0.262] | 0.080 [-0.028 to 0.209] | 0.018 [-0.089 to 0.125] | 0.141 [0.039 to 0.251]

3. Secondary Outcome: EBA Measured as the Daily Rate of Change in log10 CFUs of M. Tuberculosis in Sputum on Solid Media (Days 7-14)
Time Frame: Day 7-14
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: log10CFU/ml/day
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Number analyzed (Participants) | 13 | 12 | 15 | 13 | 15 | 14 | 15
log10CFU/ml/day | 0.085 [-0.013 to 0.175] | 0.146 [0.033 to 0.248] | 0.085 [-0.006 to 0.182] | 0.118 [-0.017 to 0.250] | 0.022 [-0.058 to 0.101] | -0.038 [-0.130 to 0.046] | 0.157 [0.048 to 0.267]

4. Secondary Outcome: EBA Expressed as the Daily Percentage Change in Time to Positive (TTP) Signal in Liquid Culture for M. Tuberculosis (Days 0-14)
Time Frame: Days 0-14
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of change in time/day
Groups:
- Clofazimine (C): clofazimine (C): 300 mg on Days 1 to 3 and 100 mg on Days 4-1414
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Number analyzed (Participants) | 13 | 14 | 15 | 13 | 15 | 14 | 15
percentage of change in time/day | 6.3 [4.2 to 8.6] | 7.0 [5.1 to 9.4] | 4.3 [2.9 to 5.7] | 4.9 [3.3 to 6.8] | 2.0 [0.8 to 3.4] | -0.3 [-1.5 to 1.0] | 6.3 [4.8 to 7.6]

5. Secondary Outcome: EBA Expressed as the Daily Percentage Change in TTP Signal in Liquid Culture for M. Tuberculosis (Day 0-2)
Time Frame: Day 0-2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of change in time/day
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Number analyzed (Participants) | 13 | 14 | 15 | 13 | 15 | 14 | 15
percentage of change in time/day | 10.6 [8.0 to 13.3] | 13.2 [9.0 to 17.9] | 6.0 [4.2 to 7.8] | 9.1 [6.5 to 12.2] | 4.7 [2.4 to 7.5] | 2.1 [-0.5 to 5.0] | 12.9 [8.9 to 17.9]

6. Secondary Outcome: EBA Expressed as the Daily Percentage Change in TTP Signal in Liquid Culture for M. Tuberculosis (Days 7-14)
Time Frame: Days 7-14
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of change in time/day
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Number analyzed (Participants) | 13 | 14 | 15 | 13 | 15 | 14 | 15
percentage of change in time/day | 3.6 [1.5 to 6.2] | 4.5 [2.9 to 6.2] | 3.1 [1.7 to 4.7] | 3.0 [1.5 to 4.9] | 0.8 [-0.7 to 2.3] | -1.3 [-2.9 to 0.4] | 4.4 [2.9 to 5.8]

ADVERSE EVENTS:
Arm/Group | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) | TMC207, PA-824 and Clofazimine (J-PA-C) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) | Pyrazinamide (Z) | Clofazimine (C) | Rifafour
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 9/15 | 8/15 | 10/15 | 10/15 | 9/15 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) (N=15) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) (N=15) | TMC207, PA-824 and Clofazimine (J-PA-C) (N=15) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) (N=15) | Pyrazinamide (Z) (N=15) | Clofazimine (C) (N=15) | Rifafour (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC207, PA-824, Pyrazinamide and Clofazimine (J-PA-Z-C) (N=15) | TMC207, PA-824 and Pyrazinamide (J-PA-Z) (N=15) | TMC207, PA-824 and Clofazimine (J-PA-C) (N=15) | TMC207, Pyrazinamide and Clofazimine (J-Z-C) (N=15) | Pyrazinamide (Z) (N=15) | Clofazimine (C) (N=15) | Rifafour (N=15)
QT prolonged (Investigations) | 3 | 0 | 3 | 2 | 1 | 0 | 0 — Electrocardiogram
ALT Increased (Investigations) | 2 | 2 | 0 | 2 | 1 | 3 | 1 — Laboratory toxicities
AST Increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 2 | 0 — Laboratory toxicities
GGT increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 — Laboratory toxicities
Transaminases increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 — Laboratory toxicities
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 — Laboratory toxicities
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Urea Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary Gland Enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 1 | 3 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1
Bundle Branch Block Right (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth Abcess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel Puncture Site Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 — and Administration site conditions
Oedema, peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 — and Administration site conditions
Foreign Body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural Dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Pressure inadequately controlled (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerumen Impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator or any Sub-Investigator shall submit any oral or written publication or abstract concerning this study to the Sponsor not less than thirty (30) days prior to submission to any journal, other publication or meeting, for review and removal of confidential information.